CLINICAL TRIAL: NCT04636619
Title: Clinical Trial Evaluating the Effect of External Evaluation and Training on the Incomplete Resection Rate in Cold Snare Polypectomies in Colonic Lesions <10 Mm (POLIPEVA Study)
Brief Title: Clinical Trial Evaluating External Evaluation and Training on the Incomplete Resection (POLIPEVA Study)
Acronym: POLIPEVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Marina de Benito Sanz, Principal Investigator, Hospital del Rio Hortega
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Colonic Polyp; Colorectal Adenoma; Colorectal Cancer
Keywords: Polypectomy,; Cold Snare polypectomy; Incomplete resection rate
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-pharmacological clinical trial evaluating the incomplete resection rate in colonic cold snare polypectomy in two phases, before and after receiving a polypectomy online course.
Masking Description: Patients are blinded to know which group their endoscopist belongs to. Pathology is blinded to know which group of endoscopists performed each polypectomy.
  A centralized research nurse, blinded to procedure and groups, will made the telephonic follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- On-line training course (Experimental): Each participant will receive the global data, the results obtained by all the endoscopists (anonymously except for each interested party, the rest being identified by codes), as well as a detailed analysis of their results, comparing them with the joint data and the 3 tertiles.
  Interventions: Procedure: Colonic polypectomy; Behavioral: Online training course

INTERVENTIONS:
Procedure: Colonic polypectomy — Cold snare resection of colorectal polyps
Behavioral: Online training course — Polypectomy technique online course

SUMMARY:
Introduction It has been shown that some quality indicators in endoscopy can be improved through educational interventions. There are marked differences in the proportion of incomplete polypectomies among endoscopists. The effectiveness of measures to improve it has not been evaluated.

Objective The main objective is to evaluate whether a training intervention or the notification of the individual proportion of incomplete polypectomies (those in which post-polypectomy biopsies of the resection margin show tissue other than normal mucosa) can improve this proportion. As secondary objectives, we will compare the proportion of fragmented polypectomies and adverse events. We will evaluate the factors associated with incomplete excision or failed cold polypectomy, as well as the individual evolution of the participants.

Methods Non-pharmacological clinical trial involving endoscopists with> 1 year of experience and patients scheduled for colonoscopy. After each polypectomy, 2 additional biopsies will be taken and evaluated centrally by a blind pathologist. In a first phase, the basal rate of the participants will be evaluated. After it, the endoscopists will receive a course on endoscopic polypectomy and the other their rate of complete resection. The number of polyps required will vary depending on the number of endoscopists The primary objective will be compared using logistic regression models based on generalized estimating equations (GEE), taking into account the within-subject correlation.

DETAILED DESCRIPTION:
Design

Non-pharmacological clinical trial

Methods

Study population The population of endoscopists under study includes specialists in the digestive system with more than one year of experience in endoscopies.

Candidate patients to be included will be those scheduled to perform a colonoscopy on a non-urgent basis. The patient will be invited to participate prior to the performance of the colonoscopy.

Stages of the study Stage I: estimation of incomplete polypectomies

All participating endoscopists will include polyps in order to perform the baseline estimate. To avoid that the estimation is made on the basis of a small group of participants, a minimum number of lesions will be required and a maximum threshold for polyps will be established. These thresholds will be estimated as follows:

Minimum: sample size / (number of participating endoscopistsx1.5). It can never be less than 25 injuries.

Maximum: sample size / (number of participating endoscopists / 1.5) Once there are a sufficient number of endoscopists who are at the thresholds allowing their samples to reach the established sample size, the end of patient recruitment will be set for the baseline estimate 30 days later. After this period, all endoscopists who do not reach the minimum threshold will be excluded from the study.

Stage II:

Online training course An online course will be offered that will explain the technique for excision of lesions with a cold loop and the importance of complete resection, techniques to determine the edges of the lesion and possible remains at the polypectomy base through images, video clips. and interaction with the speakers.

After the training measures, each endoscopist will proceed to recruit a minimum number of polyps that will be determined based on the sample size reached in phase I. Once the pre-established sample size has been reached, this phase will be closed.

E) Recruitment, procedure and follow-up Patient recruitment is the same in all phases. Patients who meet the inclusion criteria and do not present any exclusion criteria (pre-endoscopic) will be invited to participate in the study. Informed consent will be completed in accordance with law 41/2002 on patient autonomy without thereby altering the relationship with their doctor or causing any harm to their treatment.

Anonymized video clips of all polypectomies will be recorded in each of the phases, including from when the polypectomy loop is inserted into the endoscope until the biopsies are taken from the base of the polyp.

1. Endoscopic act The interventions will be carried out in each of the participating centers. The examinations will be carried out under sedation, following the protocols established in each center. Once the lesion is identified, it will be removed using a cold loop. This will be carried out following the usual standards recommended by international companies. If macroscopic remains of the lesion are observed, a fragmented polypectomy should be performed using, in the same way, the cold loop.

   Once the polypectomies are completed, its base will be carefully evaluated, taking biopsies 2 random biopsies at the base of the polypectomy, at two of the ends of the eschar.
2. Post-endoscopic follow-up In the 5th week post-colonoscopy from the endoscopic examination, the patient will be contacted by telephone to collect possible complications (they will be questioned about visits to the hospital and in a directed way about the most frequent symptoms of the usual complications (fever, bleeding, abdominal pain ), and if so, the medical history will be reviewed to assess the severity of the complication.
3. Histological analysis The analysis of the polypectomy specimens will be carried out in each center according to its usual protocol. The analysis of the biopsies of the base of the polyp will be performed centrally by a pathologist with more than 5 years of experience in digestive pathology. Samples from the base of the polyp will be sent from each center for centralized study. The pathologist will be blinded as to the histological diagnosis of the removed polyp. Samples submitted for centralized analysis will not be kept, but will be destroyed once the study is completed according to standard protocols

1) Endoscopic act The interventions will be carried out in each of the participating centers. The examinations will be carried out under sedation, following the protocols established in each center. Once the lesion is identified, it will be removed using a cold loop. This will be carried out following the usual standards recommended by international companies. If macroscopic remains of the lesion are observed, a fragmented polypectomy should be performed using, in the same way, the cold loop.

Once the polypectomies are completed, its base will be carefully evaluated, taking biopsies 2 random biopsies at the base of the polypectomy, at two of the ends of the mucosal defect.

F) Sample size According to the results obtained in our previous work, we observed an intra-subject correlation coefficient (taking the endoscopists as subjects) of 0.017.

The sample size will depend on the number of participating endoscopists. Assuming a baseline proportion of incomplete polypectomies of 7.5%, to detect an absolute risk reduction of 3.5% (that is, to identify as different proportions equal to or less than 4%) with an alpha risk of 5% and a 80% power, the required number of polyps will vary depending on the group of participating endoscopists.

According to our previous work, a 2.5% loss should also be assumed. Given that to estimate the proportion of incomplete polypectomies with a margin of error of +/- 1.5% for any value below 3.5%, a maximum of 558 polyps would be needed, in case of presenting a baseline proportion of incomplete polypectomies < 4%, we could estimate the confidence intervals accurately.

G) Data collection All the variables concerning the characteristics of the endoscopist, the patient and the injuries included will be collected in each center. The variables related to the histological diagnosis of the polypectomy specimen will be collected in the same way at the respective center. The variables concerning the follow-up will be collected centrally, through a telephone call that will be made the 5th week after the procedure. The variable related to the histological study of the base of the polyp will be collected centrally by the pathologist in charge of analyzing the samples. The video clips will be stored in a collection created de novo and centralized in the main researcher center

2) Post-endoscopic follow-up In the 5th week post-colonoscopy from the endoscopic examination, the patient will be contacted by telephone to collect possible complications (they will be questioned about visits to the hospital and in a directed way about the most frequent symptoms of the usual complications (fever, bleeding, abdominal pain ), and if so, the medical history will be reviewed to assess the severity of the complication.

3) Histological analysis The analysis of the polypectomy specimens will be carried out in each center according to its usual protocol. The analysis of the biopsies of the base of the polyp will be performed centrally by a pathologist with more than 5 years of experience in digestive pathology. Samples from the base of the polyp will be sent from each center for centralized study. The pathologist will be blinded as to the histological diagnosis of the removed polyp. Samples submitted for centralized analysis will not be kept, but will be destroyed once the study is completed according to standard protocols.

Data collection The data from the data collection notebooks will be collected anonymously by the main investigator or collaborating investigators, encrypted and dissociated from the clinical information by means of a patient identification code (ID), in a database created by the program Research Electronic Data Capture Tool (RedCap) (17) attached to the Spanish Society of Digestive Endoscopy, which allows coordinating data collection through access from different national centers. Subsequently, for their analysis, they will be merged by the principal investigator or the encrypted and dissociated collaborating investigators, in a database created using the STATA Stata Corporation program. 2013. Stata Statistical Software: Release 13. College Station, Texas: Stata Corporation. The data entered in the database will be encrypted and the database will be protected with a password to which only researchers will have access. The video clips will be completely anonymized and identified by a code, which will be provided by the main researcher. In no case will identifying data of the patient appear in said videos.

The unified file will be kept at the Río Hortega University Hospital and will be kept until the end of the study. Regarding the application of the Organic Law on Data Protection 15/1999 and the Royal Decree 1720/2007 that develops it, it should be noted that the protocol defined in the project aimed at epidemiological analysis determines that the files will record information completely anonymized.

Statistical analysis In the quantitative variables, the arithmetic mean and standard deviation will be calculated (the variables that do not follow a normal distribution according to the Kolmogorov-Smirnov test will be described with median and interquartile range), and the qualitative ones will be expressed as percentages and their intervals of 95% confidence.

The main objective, the difference in the proportion of indicators collected in the reports made with free fields or with standardized reports, will be compared using logistic regression models based on generalized estimating equations (GEE), taking into account the within-subject correlation. .

Among the secondary endpoints, the proportion of complications in both groups, the proportion of fragmented polypectomies and polypectomies that require repositioning will be compared using the homogeneity z-test without using the Yates correction. Multivariate logistic regression techniques will be used to evaluate the factors associated with incomplete polypectomies and those associated with a failed cold polypectomy. The individual evolution of the endoscopists will be displayed graphically. Cumulative summatory learning curves will be used to graphically represent the individual evolution of the endoscopists.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age scheduled for a non-urgent colonoscopy.

Exclusion Criteria:

* Absence of lesions <10 mm.
* Contraindication for polypectomy (anticoagulant treatment that cannot be withdrawn, treatment with clopidogrel, coagulopathy or severe thrombocytopenia)
* Loss of polypectomy specimen
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1920 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Incomplete resection rate | One year
  To compare the change in the proportion of incomplete cold-snare polypectomies in polyps <10mm.

CONTACTS AND LOCATIONS:
Overall Officials: Marina De Benito Sanz, MD, Principal Investigator — Hospital Río Hortega
Locations (1):
- Hospital Rio Hortega, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Ransohoff DF. Colon cancer screening in 2005: status and challenges. Gastroenterology. 2005 May;128(6):1685-95. doi: 10.1053/j.gastro.2005.04.005. No abstract available. PMID 15887159
- [Background] Baxter NN, Warren JL, Barrett MJ, Stukel TA, Doria-Rose VP. Association between colonoscopy and colorectal cancer mortality in a US cohort according to site of cancer and colonoscopist specialty. J Clin Oncol. 2012 Jul 20;30(21):2664-9. doi: 10.1200/JCO.2011.40.4772. Epub 2012 Jun 11. PMID 22689809
- [Background] Baxter NN, Goldwasser MA, Paszat LF, Saskin R, Urbach DR, Rabeneck L. Association of colonoscopy and death from colorectal cancer. Ann Intern Med. 2009 Jan 6;150(1):1-8. doi: 10.7326/0003-4819-150-1-200901060-00306. Epub 2008 Dec 15. PMID 19075198
- [Background] Mulder SA, van Soest EM, Dieleman JP, van Rossum LG, Ouwendijk RJ, van Leerdam ME, Kuipers EJ. Exposure to colorectal examinations before a colorectal cancer diagnosis: a case-control study. Eur J Gastroenterol Hepatol. 2010 Apr;22(4):437-43. doi: 10.1097/MEG.0b013e328333fc6a. PMID 19952765
- [Background] Nishihara R, Wu K, Lochhead P, Morikawa T, Liao X, Qian ZR, Inamura K, Kim SA, Kuchiba A, Yamauchi M, Imamura Y, Willett WC, Rosner BA, Fuchs CS, Giovannucci E, Ogino S, Chan AT. Long-term colorectal-cancer incidence and mortality after lower endoscopy. N Engl J Med. 2013 Sep 19;369(12):1095-105. doi: 10.1056/NEJMoa1301969. PMID 24047059
- [Background] Singh H, Nugent Z, Demers AA, Kliewer EV, Mahmud SM, Bernstein CN. The reduction in colorectal cancer mortality after colonoscopy varies by site of the cancer. Gastroenterology. 2010 Oct;139(4):1128-37. doi: 10.1053/j.gastro.2010.06.052. Epub 2010 Jun 20. PMID 20600026
- [Background] Bourke MJ. Making every colonoscopy count: Ensuring quality in endoscopy. J Gastroenterol Hepatol. 2009 Oct;24 Suppl 3:S43-50. doi: 10.1111/j.1440-1746.2009.06070.x. PMID 19799697
- [Background] Grupo de Trabajo de "Indicadores de calidad en endoscopia" de la Sociedad Espanola de Patologia Digestiva (SEPD). Quality indicators in colonoscopy. The colonoscopy procedure. Rev Esp Enferm Dig. 2018 May;110(5):316-326. doi: 10.17235/reed.2018.5408/2017. PMID 29658767
- [Background] Coe SG, Crook JE, Diehl NN, Wallace MB. An endoscopic quality improvement program improves detection of colorectal adenomas. Am J Gastroenterol. 2013 Feb;108(2):219-26; quiz 227. doi: 10.1038/ajg.2012.417. Epub 2013 Jan 8. PMID 23295274
- [Background] Ussui V, Coe S, Rizk C, Crook JE, Diehl NN, Wallace MB. Stability of increased adenoma detection at colonoscopy. Follow-up of an endoscopic quality improvement program-EQUIP-II. Am J Gastroenterol. 2015 Apr;110(4):489-96. doi: 10.1038/ajg.2014.314. Epub 2014 Sep 30. PMID 25267326
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686